CLINICAL TRIAL: NCT01675180
Title: Self Reported Oral Health, Awareness and Attitude Towards Dental Care and Risk of Dental Caries Among Pregnant Women in Norway
Brief Title: Self Reported Oral Health, Awareness and Attitude Towards Dental Care Among Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2012/633/REK nord
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy; Oral Health; Attitude; Oxidative Stress
Keywords: pregnancy, oral health, attitude, awareness, streptococcus mutans, lactobacilli, oxidative stress
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information (Other): Women randomized to the intervention will recieve information and counseling on oral health care during pregnancy
  Interventions: Other: Information; Other: Control
- Control (No Intervention)

INTERVENTIONS:
Other: Information — Women in the intervention group will recieve information and counseling on oral health care during pregnancy
  Arms: Information
Other: Control — No intervention
  Arms: Information

SUMMARY:
Purpose/Objective of the study:

The main objective of the study is to investigate oral health awareness and attitudes towards oral health among Norwegian pregnant women and assess the impact of information about oral hygiene on the risk of dental caries during pregnancy.

The hypothesis of the study are:

1. The state of oral health during pregnancy depends on pregnant woman's preventive oral hygiene behaviour and practice.
2. Pregnant women with high level of oral health awareness and positive attitude towards oral health are more likely to visit their dentists regularly and have better oral hygiene compared to those with less awareness.
3. Proper information and guidance on oral hygiene care provided during pregnancy can help to improve oral bacteriological milieu and reduce the dental caries risk among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Women with viable pregnancy ≥ 17 weeks gestation

Exclusion Criteria:

* Those not willing to participate in the study.
* Women who are unable to communicate well in Norwegian.
* Women who have been diagnosed to have a fetus with a chromosomal or structural fetal anomaly and do not plan to continue their pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Oral health | In 4 weeks interval after recrutiatment of study participants
  Streptococcus Mutans, lactobacilli

SECONDARY OUTCOMES:
Attitude | After approximately 6 months
  Attitude towards oral health care

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Acharya, Professor, Principal Investigator — University of Tromsø and University Hospital of North Norway
Locations (1):
- Department of Obstetrics and Gynaecology, University Hospital of Northern Norway (UNN), Tromsø, Troms, Norway

REFERENCES:
- [Derived] Wagle M, D'Antonio F, Reierth E, Basnet P, Trovik TA, Orsini G, Manzoli L, Acharya G. Dental caries and preterm birth: a systematic review and meta-analysis. BMJ Open. 2018 Mar 2;8(3):e018556. doi: 10.1136/bmjopen-2017-018556. PMID 29500202